CLINICAL TRIAL: NCT03018704
Title: Topiramate Treatment of Alcohol Use Disorder in African Americans
Brief Title: Topiramate Treatment of Alcohol Use Disorders in African Americans
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: In ability to recruit
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURA-010-16S
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Use Disorder
Keywords: alcoholism; treatment
MeSH Terms: conditions — Alcoholism | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): a placebo control arm
  Interventions: Drug: placebo
- Topiramate (Experimental): Topiramate an FDA approved anticonvulsant has been shown effective in the treatment of alcohol use disorder but there is no data supporting use in minority patients. The medication was dosed orally twice per day with a starting dose of 25 mg, increasing the dose as tolerated to 200mg daily in divided doses. Patient were titrated to the highest dose tolerable.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — anticonvulsant medication. The medication was dosed twice per day with a starting dose of 25 mg, increasing the dose as tolerated to 200mg daily in divided doses. Patient were titrated to the highest dose tolerable.
  Other Names: Topamax
  Arms: Topiramate
Drug: placebo — inactive medication. the doses of placebo were titrated the same as the active intervention.
  Arms: Placebo

SUMMARY:
The focus of this application is on the improvement of services for African American (AAs) Veterans afflicted with an alcohol use disorder. The project focuses on the use of topiramate as a treatment for alcohol use disorders. Despite having lower rates of heavy drinking than European Americans (EAs), AAs have significantly higher rates of mortality from a variety of alcohol-related conditions, including liver cirrhosis, accidents, and violence. Despite the higher rates of morbidity and mortality, pharmacological treatments are understudied in this population and there is some evidence that medications are less preferred and less effective in AAs.

DETAILED DESCRIPTION:
1. Objective(s): Despite having lower rates of drinking and heavy drinking than European Americans (EAs), African Americans (AA) have significantly higher rates of mortality from a variety of alcohol-related conditions, including liver cirrhosis, accidents, and violence. The current proposal aims to improve alcohol treatment in AA Veterans, who comprise 12% of the Veteran population.
2. Research Design: The proposed study is a two-arm, randomized 12-week, parallel-groups comparison of topiramate versus placebo to reduce the frequency of heavy drinking days and increase the number of abstinent days in 160 AA patients with AUD.
3. Methodology: The following specific aim is used to direct the methods:

   Specific Aim 1. Understanding health disparities. Aim 1 will focus on the screening process, using the screening outcomes data, including reasons for patients declining to participate in the trial, to conduct descriptive analyses of the screening process and recruitment efforts. We will supplement this description by examining changes in drinking and motivation for treatment before and during the pandemic. In the resultant manuscript, we will also discuss strategies for recruiting a minority population to participate in addiction treatment studies.

   Specific Aim 2. Future study planning with safety results. Aim 2 will focus on assessing the safety and tolerability of topiramate dosing, which will provide the basis for evaluating the risks associated with topiramate treatment for reducing heavy drinking in AAs. The additional participants will greatly improve our effect size estimate, pooling across sites; for example, the width of a confidence interval on a difference in means at the end of the study based on a sample of size 80 will be 61% of the width of a corresponding confidence interval based on a sample of size 30. In addition, two sites will also provide information on treatment-by-site heterogeneity, which will be useful for informing the design of a multi-site trial, which we believe is the best option for recruiting an adequate sample for a well powered efficacy trial. To increase the number of subjects exposed to topiramate treatment, we will randomize participants to a 2:1 ratio of topiramate to placebo treatment.

   Specific Aim 3. Combined analysis with available RCT datasets. We have data available from two completed RCTs of topiramate that used a design almost identical to that of the present study (n's = 138 and 170, including 16 AAs). We plan to conduct an analysis that combines the data from the three trials, to test for differences in efficacy by population group (i.e., AAs and EAs), and to compare adverse event profiles across population groups. Combining the datasets will allow analyses that incorporate individual-level heterogeneity, in contrast to meta-analyses, where typically only group comparisons would be possible. This will be accomplished using de-identified data from each study.
4. Impact/Significance: The proposal is innovative in that it will focus on AAs with AUD, an understudied and underserved population for whom no such data currently exist. Given the far-reaching effects of AUD and its high prevalence among Veterans, added evidence based treatments may realize reduced health care costs from unnecessary ED visits and reduced complications of illnesses such as hepatitis C and congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. self-identification as African American;
2. age 18 to 70 years, inclusive;
3. average weekly ethanol consumption of >24 standard drinks for men or >18 standard drinks for women, with a weekly average of > 2 heavy drinking days (men: > 5 standard drinks; women: > 4 standard drinks) during the month before screening;
4. a current diagnosis of moderate or severe AUD (i.e., meeting at least 4 of 11 DSM-5 AUD criteria);
5. expressed goal to reduce or stop drinking;
6. able to read English at the 6th grade or higher level and without gross cognitive impairment;
7. women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or are less than two years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative urine pregnancy test prior to initiation of treatment
8. willing and able to provide signed, informed consent to participate in the study.

Exclusion Criteria:

1. a current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including direct bilirubin elevations of >110% or a transaminase elevation >300% of normal;
2. history of nephrolithiasis;
3. history of glaucoma;
4. current serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, antisocial personality disorder, or imminent suicide or violence risk);
5. current moderate-to-severe alcohol withdrawal requiring pharmacological treatment (see Section D.4.a. regarding alcohol detoxification);
6. current DSM-IV diagnosis of drug use disorder (other than nicotine or cannabis) or a urine drug screen positive for recent use of opioids, cocaine, or amphetamines (may be repeated once and if the result is negative on repeat it is not exclusionary);
7. a history of hypersensitivity to TOP;
8. current regular treatment with more than one antidepressant or any treatment with a tricyclic antidepressant;
9. current treatment with a psychotropic medication (with the exception of antidepressants where monotherapy is allowable), including medications that, when combined with alcohol or TOP, present a risk of overdose or significant adverse effect (e.g., chronic opioid use) (of note we will allow subjects to discontinue medications that have no demonstrated therapeutic effect in order to enroll - amount of time off of the medication will be a clinical decision left to the discretion of the study physician investigators);
10. current treatment with TOP or a medication approved for AUD;
11. considered to be unsuitable candidates for receipt of an investigational drug;
12. treatment with carbonic anhydrase inhibitors, due to the added risk of metabolic acidosis,
13. Body Mass Index (BMI) of less than 18.5.
14. untreated gout as topiramate has been shown in one study to increase uric acid.
15. current treatment with dolutegravir.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from VA outpatient and inpatient mental health and addiction programs. Recruitment occurred between October 2017 through May 2020
Pre-assignment Details: Prior to randomization, consented individuals (n=79) were assessed for participation. The majority of non randomized subjects (n=31) didn't meet inclusion criteria (not drinking) or exclusion criteria (other drugs). I addition 5 subjects withdrew consent before randomization and 6 were lost to follow up. That lead to 37 who were randomized.
Groups:
- Placebo: a placebo control arm
  placebo: inactive medication
- Topiramate: Topiramate an FDA approved anticonvulsant has been shown effective in the treatment of alcohol use disorder but there is no data supporting use in minority patients.
  Topiramate: anticonvulsant medication
Period: Overall Study
Arm/Group | Placebo | Topiramate
Started | 19 | 18
Completed | 18 | 17
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Topiramate | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10.2) | 48 (11.6) | 49.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37
Percent Heavy Drinking days [Mean (Standard Deviation); unit: percent of trial days of heavy drinking] — Drinking was recorded using the timeline follow back methodology which is an interview based method to record drinking on each day. The summary measure counts the number of days of heavy drinking (>4drinks per day) divided by the number of observation days to report the percent of observation days for which there is heavy drinking. For the prestudy period, the observation period is 90 days.
  percent of trial days of heavy drinking | 70.8 (20.4) | 62.8 (23.4) | 67 (22)
Depression rating (PHQ9) [Mean (Standard Deviation); unit: units on a scale] — Depression scale range 0-27 higher indicates more depression
  units on a scale | 8.6 (7.6) | 11.4 (7.0) | 10. (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent Days of Heavy Drinking
Description: Drinking was recorded using the timeline follow back methodology which is an interview based method to record drinking on each day during the trial. The summary measure (% days heavy drinking) counts the number of days of heavy drinking (>4drinks per day) divided by the number of observation days to report the percent of observation days for which there is heavy drinking. For the the outcome measure the observation period is the last 42 days of the trial.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days of heavy drinking
Arm/Group | Placebo | Topiramate
Number analyzed (Participants) | 18 | 17
percentage of days of heavy drinking | 26.7 (24.9) | 14.8 (14.6)

ADVERSE EVENTS:
Time Frame: Adverse events are measured at each study visit during the trial and reported as a summary of events over the 12 weeks.
Description: No difference
Arm/Group | Placebo | Topiramate
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

LIMITATIONS AND CAVEATS:
The study was stopped by the funding agency due to difficulty recruiting during COVID pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03018704/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03018704/ICF_001.pdf